CLINICAL TRIAL: NCT06859710
Title: Interactions Between Delta-9-THC and CBD: A Controlled Human Drug-administration Study Probing a Harm Reduction Strategy
Brief Title: THC and CBD: A Controlled Human Study Probing a Harm Reduction Strategy
Acronym: THC-REDUX
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Ziva D. Cooper, PhD, Professor, University of California, Los Angeles
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 24-5306; 93306 (Other Grant/Funding Number: CA Department of Cannabis Control)
Record Dates: First submitted 2025-02-25; First posted 2025-03-05 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-09

CONDITIONS: Abuse, Drug; Pain
Keywords: Cannabis; THC; CBD
MeSH Terms: conditions — Substance-Related Disorders; Pain; Marijuana Abuse | interventions — nabiximols; Dronabinol

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blind, placebo-controlled study. All participants will complete all dose conditions in a randomized order.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Placebo (Placebo Comparator): 0 mg THC, 0 mg CBD
  Interventions: Drug: Placebo
- THC (Active Comparator): 20 mg THC, 0 mg CBD
  Interventions: Drug: THC
- CBD 20 (Active Comparator): 0 mg THC, 20 mg CBD
  Interventions: Drug: CBD 20 mg
- CBD 40 (Active Comparator): 0 mg THC, 40 mg CBD
  Interventions: Drug: CBD 40 mg
- CBD 80 (Active Comparator): 0 mg THC, 80 mg CBD
  Interventions: Drug: CBD 80 mg
- THC with CBD 20 (Active Comparator): 20 mg THC, 20 mg CBD
  Interventions: Drug: THC; Drug: CBD 20 mg
- THC with CBD 40 (Active Comparator): 20 mg THC, 40 mg CBD
  Interventions: Drug: THC; Drug: CBD 40 mg
- THC with CBD 80 (Active Comparator): 20 mg THC, 80 mg CBD
  Interventions: Drug: THC; Drug: CBD 80 mg

INTERVENTIONS:
Drug: Placebo — Vaporized Placebo
  Other Names: Cannabis
  Arms: Placebo
Drug: THC — Vaporized THC (20 mg)
  Other Names: Cannabis
  Arms: THC; THC with CBD 20; THC with CBD 40; THC with CBD 80
Drug: CBD 20 mg — Vaporized CBD (20 mg)
  Other Names: Cannabis
  Arms: CBD 20; THC with CBD 20
Drug: CBD 40 mg — Vaporized CBD (40 mg)
  Other Names: Cannabis
  Arms: CBD 40; THC with CBD 40
Drug: CBD 80 mg — Vaporized CBD (80 mg)
  Other Names: Cannabis
  Arms: CBD 80; THC with CBD 80

SUMMARY:
The purpose of this research is to assess the impact of CBD on the effects of THC.

DETAILED DESCRIPTION:
Some evidence indicates that cannabidiol (CBD), a non-intoxicating cannabis component, might mitigate certain effects of THC. This study will examine possible roles for CBD in modulating THC's adverse and analgesic effects.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant and non-lactating females aged 21-55 years
* Report cannabis use 1-7 days per week over the month prior to screening
* Not currently seeking treatment for their cannabis use
* History of inhaled cannabis use
* Have a Body Mass Index from 18.5 - 34 kg/m2
* Able to perform all study procedures
* Must be using a contraceptive (hormonal or barrier methods)

Exclusion Criteria:

* Meeting DSM-V criteria for severe Cannabis Use disorder (CUD) or any substance use disorder other than nicotine, caffeine, mild or moderate CUD
* Evidence of severe psychiatric illness (e.g. mood or anxiety disorder with functional impairment or suicide risk, schizophrenia) judged by the study physician (and PI) to put the participant at greater risk of experiencing adverse events due to completion of study procedures, interfere with their ability to participate in the study, or their capacity to provide informed consent.
* Report using other illicit drugs in the prior 4 weeks
* Current pain
* Pregnancy
* Currently enrolled in another research protocol
* Not using a contraceptive method (hormonal or barrier methods)
* Insensitivity to the cold water stimulus of the Cold Pressor Test
* Any disorders that might make cannabis administration hazardous as determined by evaluation physician after review of all medical assessments along with medical history.
* Not able to speak and read English

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-11-05 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Subject-rated drug effects of abuse liability | 3 hours
  Subject ratings of "Good Drug Effect" as measured using a visual analog scale (1-100 mm)
Analgesia as measured using the Cold Pressor Test | 3 hours
  Pain threshold assessed using the Cold Pressor Test (percent baseline)
Behavioral task performance as assessed by the DRUID App Score | 3 hours
  Trough composite scores on the DRUID App
Pharmacokinetics of THC | 3 hours
  Peak plasma levels of THC (ng/ml)

CONTACTS AND LOCATIONS:
Overall Officials: Ziva Cooper, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Center for Cannabis and Cannabinoids, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No